CLINICAL TRIAL: NCT06418685
Title: The First Affiliated Hospital of Naval Medical University
Brief Title: Real-World Clinical Study on the Efficacy of Vibrating Capsule (Vibrabot Capsule) for Chronic Functional Constipation
Acronym: RWS-VC
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Ruijin Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Shanghai 10th People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai 6th People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Pudong New Area Gongli Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ANKONYX2023006
Record Dates: First submitted 2024-01-30; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-01

CONDITIONS: Clinical Study; Chronic Functional Constipation
Keywords: Real-World Clinical Study; Vibrating Capsule; Chronic Functional Constipation; Response Rate; Complete Spontaneous Bowel Movement
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VC group: Treatment with Vibrabot Capsule
  Interventions: Device: Treatment with Vibrating Capsule
- Other treatment group: Selecting Alternative Treatment Methods through Assessment

INTERVENTIONS:
Device: Treatment with Vibrating Capsule — Main parameters of Vibrabot capsule: nominal diameter: 11.8±1mm; nominal length: 26.7±1mm; nominal weight: 4.5±1g.
  After the patient swallows the Vibrabot capsule, the capsule runs through the stomach → duodenum → jejunum and ileum → colon. According to the clinical data and configuration settings, the capsule will reach the colon and vibrate 8 hours after activation for ≥ 180 minutes in a cycle at low, medium, and high frequencies sequentially. The capsule relieves and treats constipation by massaging the colon wall through motor vibration to relieve colon muscle spasms and promote colonic peristalsis.
  The VC well be taken between 21:00 and 22:00 every day, and the frequency of administration is determined based on the patient's individual situation.
  Groups: VC group

SUMMARY:
This study is a multi-center prospective cohort study, which plans to include 300 patients with chronic functional constipation to treat with Vibrabot capsules, and at the same time, include ≥300 patients receiving constipation treatment during the same period.

During the study, it is necessary to collect the patients' basic information, baseline constipation status and treatment information, capsule intake during treatment, and concomitant medication. During the treatment phase, patients follow the doctor's advice to receive Vibrabot capsule treatment and maintain stable dietary intake and exercise according to the constipation diagnosis and treatment guidelines.

During the study, patients need to scan the two-dimensional code or search for the electronic questionnaire "Vibrabot Health" Official Account on WeChat, and fill in the relevant information during the treatment in the electronic questionnaire in a timely and truthful manner. The treatment effect of the patients is evaluated by assessing the number of occurrences of spontaneous bowel movements (SBM) and complete spontaneous bowel movements (CSBM).

DETAILED DESCRIPTION:
Constipation is characterized by a decrease in bowel movements, dry and hard stools, and difficulty in defecation. With changes in diet, faster pace of life, and social psychological factors, the prevalence of chronic constipation is on the rise. The global incidence of chronic constipation is 14%, while the prevalence of chronic constipation in adults in China is 4.0% to 10.0%. The prevalence of functional constipation in China is 6%. The high-risk groups for constipation include the elderly, women, diabetics, those taking opiates, antipsychotic drugs, or bedridden patients. Occupation, lifestyle, dietary habits, mental health, family history of constipation, and BMI are factors related to constipation.

Constipation affects patients' quality of life, and some patients abuse laxatives or repeatedly seek medical treatment, increasing medical costs. The main treatments for constipation are adjusting lifestyle, medication, psychotherapy, biofeedback, and surgery. However, these methods often have side effects, and patient satisfaction is still relatively low. A new approach needs to be explored to address this clinical problem.

The Disposable Gastrointestinal Vibrating Capsule System (Vibrabot capsule) (NMPA Device Approval No. 20223090282) is the world's first approved and marketed product for treating constipation through purely physical means. It can provide intermittent comfortable massages to the digestive tract, activate the intestinal neural network, awaken intestinal motility, and help alleviate constipation issues. Clinical study results show that the product is safe to use and can increase the frequency of bowel movements in patients with chronic functional constipation.

This study focuses on post-marketing clinical study for patients with functional constipation of varying severity, further evaluating the efficacy of the product in a large sample population.

Through this real-world study, to analyze the response of functional constipation patients with different severity, treatment status, capsule dosage, and combined medication to Vibrabot capsule, as well as the duration of efficacy maintenance during the follow-up period; to compare the efficacy with patients treated with drugs or other therapies during the same period, explore the possibility of curing functional constipation patients, further improve the treatment satisfaction of constipation patients, and promote the establishment and application of consensus or guidelines for the use of Vibrabot capsule in treating functional constipation.

Each patient will undergo a series of study visits, including screening, treatment visit, and follow-up visit. The visit process is briefly described as follows:

Visit 1 (0 ~ 1 day) - Baseline/Screening Period:

This visit includes:

The patient will sign an informed consent form; Set the inclusion/exclusion criteria; Guide patients to fill out the questionnaire using the Official Account and complete the Baseline Period Questionnaire in the Official Account.

Prescription Vibrabot capsule treatment or other treatment options.

Visit 2 (Week 2 ±3 days) - Treatment Period 1:

This visit includes:

Fill out the Daily Bowel Movement Questionnaire in the WeChat Official Account every day, take Vibrabot capsules on time or opt for other treatment plans; Fill out the Constipation Symptom Self-Assessment Scale and Assessment Scale for Quality of Life with Constipation in the Official Account every 2 treatment weeks.

Record adverse events and concomitant treatments; Prescription Vibrabot capsules or other treatment options. Visit 3 (Week 4±3 days) - Treatment Period 2

This visit includes:

Fill out the Daily Bowel Movement Questionnaire in the WeChat Official Account every day, take Vibrabot capsules on time or opt for other treatment plans; Fill out the Constipation Symptom Self-Assessment Scale and Assessment Scale for Quality of Life with Constipation in the Official Account every 2 treatment weeks.

Record adverse events and concomitant treatments; Prescription Vibrabot capsules or other treatment options. Visit 4 (Week 6 ±3 days) - Treatment Period 3

This visit includes:

Fill out the Daily Bowel Movement Questionnaire in the WeChat Official Account every day, take Vibrabot capsules on time or opt for other treatment plans; Fill out the Constipation Symptom Self-Assessment Scale and Assessment Scale for Quality of Life with Constipation in the Official Account every 2 treatment weeks.

Record adverse events and concomitant treatments.

Visit 5 (Week 10±3 days) - Follow-up Period:

This visit includes:

Fill out the Daily Bowel Movement Questionnaire in the WeChat Official Account every day; Fill out the Constipation Symptom Self-Assessment Scale and Assessment Scale for Quality of Life with Constipation in the Official Account every 2 treatment weeks; Record adverse events and concomitant treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who can be diagnosed with functional constipation according to the Rome IV criteria.
2. Patients who consent to participate in this trial and voluntarily sign the informed consent form (ICF).

Exclusion Criteria:

1. People who are not eligible for surgery or refuse to undergo any abdominal surgery;
2. People with known or suspected gastrointestinal obstruction, stenosis, diverticulum, bleeding, malformation, and fistula.
3. People allergic to polymeric materials;
4. People implanted with cardiac pacemakers and using gastrointestinal pacemakers;
5. People with abdominal aortic aneurysms, gastrointestinal vascular lesions, ulcers, and lesions with bleeding tendencies.
6. People with dysphagia;
7. Pregnant women;
8. People with severe depression and anxiety and severe acute gastrointestinal lesions.
9. People with other conditions, so the investigator considers them not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multi-center clinical trial. Patients are considered eligible for this study if they meet the inclusion criteria and do not meet any of the exclusion criteria. This study plans to include 300 patients with chronic functional constipation to treat with Vibrabot capsules for at least 6 weeks, and ≥300 patients with constipation receiving other treatments concurrently.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
After treatment, whether the response rate of patients using the Vibrabot vibrating capsules alone reaches 50%. | At the end of the sixth week of treatment
  The definition of the responder is a patient with an average weekly increase of ≥1 complete spontaneous bowel movement (CSBM) compared to the baseline.

SECONDARY OUTCOMES:
Proportion of constipated patients who use/do not use other constipation treatment methods | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires.
Proportion of constipated patients who use/do not use other constipation treatment methods | at the end of the 4-week follow-up
  Collect relevant data through daily defecation questionnaires.
Proportion of patients with an average increase of ≥1 CSBMs per week compared to the baseline period | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires,CSBM refers to spontaneous defecation without anal obstruction and without taking laxatives within 24 hours before defecation.
Proportion of respondents with an average of ≥3 SBMs per week during the treatment period | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires, SBM refers to spontaneous defecation without taking laxatives within 24 hours before defecation.
Proportion of subjects with ≥3 SBMs per week and an increase of ≥1 CSBMs during at least 4 weeks of treatment compared to baseline | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires, SBM refers to spontaneous defecation without taking laxatives within 24 hours before defecation.CSBM refers to spontaneous defecation without anal obstruction and without taking laxatives within 24 hours before defecation.
Proportion of patients with an average increase of ≥1 CSBMs per week during the follow-up phase compared to the baseline period; | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires.
Proportion of patients with an average of ≥3 SBMs per week during the follow-up phase | at the end of the 4-week follow-up
  Collect relevant data through daily defecation questionnaires.
Proportion of patients with a reduction of ≥1 point in total Patient Assessment of Constipation Quality of Life questionnaire(PAC-QOL) scores after treatment compared to the baseline period | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires. Patient Assessment of Constipation Quality of Life questionnaire，The PAC-QoL questionnaire consists of 28 items, each with a score of 0 to 4, measuring anxiety, physical discomfort, psychosocial discomfort, and treatment satisfaction, respectively The higher the score, the worse the quality of life.
Proportion of patients with a reduction of ≥1 point in total Patient Assessment of Constipation Symptom (PAC-SYM) scores after treatment compared to the baseline period | At the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires.The PAC-SYM questionnaire consists of 12 items, each with a score of 0 to 4, quantifying stool symptoms, rectal symptoms, and abdominal symptoms. The higher the score, the more constipation symptoms will be serious.
Time of first use of laxative or enema after a course of vibrating capsule treatment (6 weeks) | After the end of the sixth week of treatment
  Collect relevant data through daily defecation questionnaires.

OTHER OUTCOMES:
Proportion of constipated patients (including different constipation types, occupations, age groups, BMI, gender, and baseline treatment status) responding to vibrating capsule treatment. | At the end of the sixth week of treatment
  Collect relevant data through baseline questionnaire.
occupations, age groups, BMI, gender, and baseline treatment status) responding to vibrating capsule treatment. | at the end of the 4-week follow-up period.
  Collect relevant data through baseline questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD, Study Chair — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scott SM, Simren M, Farmer AD, Dinning PG, Carrington EV, Benninga MA, Burgell RE, Dimidi E, Fikree A, Ford AC, Fox M, Hoad CL, Knowles CH, Krogh K, Nugent K, Remes-Troche JM, Whelan K, Corsetti M. Chronic constipation in adults: Contemporary perspectives and clinical challenges. 1: Epidemiology, diagnosis, clinical associations, pathophysiology and investigation. Neurogastroenterol Motil. 2021 Jun;33(6):e14050. doi: 10.1111/nmo.14050. Epub 2020 Dec 2. PMID 33263938
- [Background] Zhu JH, Qian YY, Pan J, He C, Lan Y, Chen WN, Wang BM, Zhao W, Li JN, Li XQ, Lv B, Fan YH, Zuo XL, Li Z, Zou DW, Li ZS, Liao Z. Efficacy and safety of vibrating capsule for functional constipation (VICONS): A randomised, double-blind, placebo-controlled, multicenter trial. EClinicalMedicine. 2022 Apr 25;47:101407. doi: 10.1016/j.eclinm.2022.101407. eCollection 2022 May. PMID 35518121
- [Background] Camilleri M, Kerstens R, Rykx A, Vandeplassche L. A placebo-controlled trial of prucalopride for severe chronic constipation. N Engl J Med. 2008 May 29;358(22):2344-54. doi: 10.1056/NEJMoa0800670. PMID 18509121

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT06418685/Prot_SAP_000.pdf